CLINICAL TRIAL: NCT02163577
Title: A Randomized, Open-Label, Dose Finding, Phase 2 Study to Assess the Pharmacodynamics and Safety of the Anti-FGF23 Antibody, KRN23, in Pediatric Patients With X-linked Hypophosphatemia (XLH)
Brief Title: Study of KRN23 (Burosumab), a Recombinant Fully Human Monoclonal Antibody Against Fibroblast Growth Factor 23 (FGF23), in Pediatric Subjects With X-linked Hypophosphatemia (XLH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UX023-CL201
Expanded Access: NCT03775187 (Available)
Record Dates: First submitted 2014-06-09; First posted 2014-06-13 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: X-linked Hypophosphatemia
Keywords: X-linked hypophosphatemia; XLH; FGF23; KRN23
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — burosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Burosumab Q2W (Experimental): Burosumab subcutaneous (SC) injections every 2 weeks (Q2W). Dose was determined by the participant's weight and prescribed dose by their study doctor.
  Interventions: Biological: burosumab
- Burosumab Q4W Then Q2W (Experimental): Burosumab SC injections every 4 weeks (Q4W). Dose was determined by the participant's weight and prescribed dose by their study doctor. Participants in Q4W were to switch to Q2W beginning with Week 64 dosing.
  Interventions: Biological: burosumab

INTERVENTIONS:
Biological: burosumab — solution for SC injection
  Other Names: KRN23; Crysvita®; UX023

SUMMARY:
The objectives of the study are to:

* Identify a dose and dosing regimen of burosumab, based on safety and pharmacodynamic (PD) effect, in pediatric XLH participants
* Establish the safety profile of burosumab for the treatment of children with XLH including ectopic mineralization risk, cardiovascular effects, and immunogenicity profile
* Characterize the pharmacokinetic (PK)/PD profile of the KRN23 doses tested in the monthly (Q4) and biweekly (Q2) dose regimens in pediatric XLH patients
* Determine the PD effects of burosumab treatment on markers of bone health in pediatric XLH patients
* Obtain a preliminary assessment of the clinical effects of burosumab on bone health and deformity, muscle strength, and motor function
* Obtain a preliminary assessment of the effects of burosumab on participant-reported outcomes, including pain, disability, and quality of life in pediatric XLH patients
* Evaluate the long-term safety and efficacy of burosumab

ELIGIBILITY:
Inclusion

1. Male or female, aged 5 - 12 years, inclusive, with open growth plates
2. Tanner stage of 2 or less based on breast and testicular development
3. Diagnosis of XLH supported by ONE of the following:

   * Confirmed Phosphate regulating gene with homology to endopeptidases located on the X chromosome (PHEX) mutation in the patient or a directly related family member with appropriate X-linked inheritance
   * Serum FGF23 level > 30 pg/mL by Kainos assay
4. Biochemical findings associated with XLH including:

   * Serum phosphorus ≤ 2.8 mg/dL (0.904 mmol/L)*
   * Serum creatinine within age-adjusted normal range*
5. Standing height < 50th percentile for age and gender using local normative data.
6. Radiographic evidence of active bone disease including rickets in the wrists and/or knees, AND/OR femoral/tibial bowing, OR, for expansion subjects, a Rickets Severity Score (RSS) score in the knee of at least 1.5 as determined by central read.
7. Willing to provide access to prior medical records for the collection of historical growth, biochemical and radiographic data, and disease history.
8. Provide written or verbal assent (if possible) and written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures.
9. Must, in the opinion of the investigator, be willing and able to complete all aspects of the study, adhere to the study visit schedule and comply with the assessments.
10. Females who have reached menarche must have a negative pregnancy test at Screening and undergo additional pregnancy testing during the study. If sexually active, male and female subjects must be willing to use an acceptable method of contraception for the duration of the study.

    * Criteria to be determined based on overnight fasting (minimum 4 hours) values collected at Screening Visit 2

Exclusion

1. Use of a pharmacologic vitamin D metabolite or analog (e.g. calcitriol, doxercalciferol, alfacalcidiol, and paricalcitol) within 14 days prior to Screening Visit 2; washout will take place during the Screening Period
2. Use of oral phosphate within 7 days prior to Screening Visit 2; washout will take place during the Screening Period
3. Use of calcimimetics, aluminum hydroxide antacids (e.g. Maalox® and Mylanta®), systemic corticosteroids, and thiazides within 7 days prior to Screening Visit 1
4. Use of growth hormone therapy within 3 months before Screening Visit 1
5. Use of bisphosphonates for 6 months or more in the 2 years prior to Screening Visit 1
6. Presence of nephrocalcinosis on renal ultrasound graded ≥ 3 based on the following scale: 0 = Normal 1 = Faint hyperechogenic rim around the medullary pyramids 2 = More intense echogenic rim with echoes faintly filling the entire pyramid 3 = Uniformly intense echoes throughout the pyramid 4 = Stone formation: solitary focus of echoes at the tip of the pyramid
7. Planned or recommended orthopedic surgery, including staples, 8-plates or osteotomy, within the clinical trial period
8. Hypocalcemia or hypercalcemia, defined as serum calcium levels outside the age-adjusted normal limits *
9. Evidence of tertiary hyperparathyroidism as determined by the Investigator
10. Use of medication to suppress parathyroid hormone (PTH) (e.g. Sensipar®, cinacalcet, calcimimetics) within 2 months prior to Screening Visit 1
11. Presence or history of any condition that, in the view of the investigator, places the subject at high risk of poor treatment compliance or of not completing the study
12. Presence of a concurrent disease or condition that would interfere with study participation or affect safety
13. Previously diagnosed with human immunodeficiency virus antibody, hepatitis B surface antigen, and/or hepatitis C antibody
14. History of recurrent infection or predisposition to infection, or of known immunodeficiency
15. Use of a therapeutic monoclonal antibody within 90 days prior to Screening Visit 1 or history of allergic or anaphylactic reactions to any monoclonal antibody
16. Presence or history of any hypersensitivity to recombinant human immunoglobulin G1 (IgG1) monoclonal antibody to FGF23 (burosumab) excipients that, in the judgment of the investigator, places the subject at increased risk for adverse effects
17. Use of any investigational product or investigational medical device within 30 days prior to screening, or requirement for any investigational agent prior to completion of all scheduled study assessments

    * Criteria to be determined based on overnight fasting (minimum 4 hours) values collected at Screening Visit 2

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2014-07-02 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (9):
- United States (4):
  - University of California San Francisco, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Indiana University Hospital, Indianapolis, Indiana
  - Shriners Hospital for Children, St Louis, Missouri
- Bicetre Hospital, Le Kremlin-Bicêtre, France
- University Medical Center Groningen, Groningen, Netherlands
- United Kingdom (3):
  - Royal Manchester Hospital, Manchester, Lancashire
  - Birmingham Children's University, Birmingham
  - Great Ormond Street Hospital, London

REFERENCES:
- [Derived] Linglart A, Imel EA, Whyte MP, Portale AA, Hogler W, Boot AM, Padidela R, Van't Hoff W, Gottesman GS, Chen A, Skrinar A, Scott Roberts M, Carpenter TO. Sustained Efficacy and Safety of Burosumab, a Monoclonal Antibody to FGF23, in Children With X-Linked Hypophosphatemia. J Clin Endocrinol Metab. 2022 Feb 17;107(3):813-824. doi: 10.1210/clinem/dgab729. PMID 34636899
- [Derived] Mao M, Carpenter TO, Whyte MP, Skrinar A, Chen CY, San Martin J, Rogol AD. Growth Curves for Children with X-linked Hypophosphatemia. J Clin Endocrinol Metab. 2020 Oct 1;105(10):3243-9. doi: 10.1210/clinem/dgaa495. PMID 32721016
- [Derived] Carpenter TO, Whyte MP, Imel EA, Boot AM, Hogler W, Linglart A, Padidela R, Van't Hoff W, Mao M, Chen CY, Skrinar A, Kakkis E, San Martin J, Portale AA. Burosumab Therapy in Children with X-Linked Hypophosphatemia. N Engl J Med. 2018 May 24;378(21):1987-1998. doi: 10.1056/NEJMoa1714641. PMID 29791829

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Burosumab Q2W: Burosumab SC injections every 2 weeks (Q2W). Dose is determined by the participant's weight and prescribed dose by their study doctor.
- Burosumab Q4W Then Q2W: Burosumab subcutaneous (SC) injections every 4 weeks (Q4W). Dose is determined by the participant's weight and prescribed dose by their study doctor. Participants in Q4W were to switch to Q2W beginning with Week 64 dosing.
- Total: Total of all reporting groups
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.7 (1.72) | 8.3 (2.04) | 8.5 (1.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 12 | 12 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 0 | 2
  White | 23 | 23 | 46
  Other, Not Specified | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 26 | 24 | 50
Rickets Severity Score (RSS) Total Score [Mean (Standard Deviation); unit: score on a scale] — The RSS system is a 10-point radiographic scoring method that was developed to assess the severity of nutritional rickets in the wrists and knees based on the degree of metaphyseal fraying, cupping, and the proportion of the growth plate affected. Scores are assigned for the unilateral wrist and knee X-rays deemed by the rater to be the more severe of the bilateral images. The maximum total score on the RSS is 10 points and the minimum score is 0, with a total possible score of 4 points for the wrists and 6 points for the knees. Higher scores indicate greater rickets severity.
  score on a scale | 1.92 (1.172) | 1.67 (0.999) | 1.80 (1.086)
Serum Phosphorus [Mean (Standard Deviation); unit: mg/dL] | 2.38 (0.405) | 2.28 (0.299) | 2.33 (0.356)
Serum 1, 25-Dihydroxyvitamin D [Mean (Standard Deviation); unit: pg/mL] | 41.28 (21.967) | 41.37 (15.293) | 41.33 (18.740)
Ratio of Renal Tubular Maximum Reabsorption Rate of Phosphate to Glomerular Filtration Rate(TmP/GFR) [Mean (Standard Deviation); unit: mg/dL] — Data for urinary phosphorus and tubular reabsorption of phosphate (TRP) were used in the calculation of TmP/GFR. Population: participants with a Baseline measurement
  mg/dL
    number analyzed (Participants) | 25 | 25 | 50
    (all) | 2.176 (0.4925) | 1.978 (0.3474) | 2.077 (0.4335)
RSS Knee and Wrist Scores [Mean (Standard Deviation); unit: score on a scale] — The RSS system is a 10-point radiographic scoring method that was developed to assess the severity of nutritional rickets in the wrists and knees based on the degree of metaphyseal fraying, cupping, and the proportion of the growth plate affected. Scores are assigned for the unilateral wrist and knee X-rays deemed by the rater to be the more severe of the bilateral images. The maximum total score on the RSS is 10 points and the minimum score is 0, with a total possible score of 4 points for the wrists and 6 points for the knees. Higher scores indicate greater rickets severity.
  score on a scale
    Knee Score | 1.21 (0.681) | 1.19 (0.601) | 1.20 (0.636)
    Wrist Score | 0.71 (0.619) | 0.48 (0.519) | 0.60 (0.578)
Growth Velocity [Mean (Standard Deviation); unit: cm/year] — Baseline growth velocity was calculated based on the standing height measured within 2 years prior to Baseline. Population: Data presented for participants with evaluable growth velocity data at Baseline. Growth velocity could not be calculated for 3 participants for whom pretreatment height data were not available within 2 years prior to Baseline.
  cm/year
    number analyzed (Participants) | 25 | 24 | 49
    (all) | 5.45 (1.171) | 5.24 (1.402) | 5.35 (1.280)
Standing Height Z-Score [Mean (Standard Deviation); unit: Z score] — Standing height Z scores are measures of height adjusted for a child's age and sex. The Z score indicates the number of standard deviations away from a reference population (from the Centers for Disease Control [CDC] growth charts) in the same age range and with the same sex. A Z score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z scores indicate a better outcome
  Z score | -1.72 (1.026) | -2.05 (0.957) | -1.89 (0.996)
Growth (Standing Height, Sitting Height, Arm Length, Leg Length) [Mean (Standard Deviation); unit: cm]
  Standing Height | 123.28 (10.326) | 119.42 (12.623) | 121.35 (11.584)
  Sitting Height | 70.10 (5.632) | 67.04 (5.691) | 68.57 (5.815)
  Arm Length | 54.80 (4.930) | 52.59 (6.129) | 53.70 (5.619)
  Leg Length | 66.06 (7.027) | 63.71 (8.322) | 64.89 (7.718)
6-Minute Walk Test (6MWT) Distance (Predicted Percent of Normal) [Mean (Standard Deviation); unit: percentage of predicted distance] — The total distance walked (meters) in a 6-minute period was measured. The percent of predicted values were calculated using published normative data based on age, gender, and height (Geiger et al. 2007).
  percentage of predicted distance | 79.32 (13.257) | 81.42 (15.101) | 80.37 (14.109)
POSNA-PODCI Normative Scores [Mean (Standard Deviation); unit: T-score] — The Pediatric Orthopedic Society of North America Pediatric Outcomes Data Collection Instrument (POSNA-PODCI) yields 4 functional assessment scores: Upper Extremity Function,Transfers and Basic Mobility, Sports/Physical Function, and Comfort/Pain. Also a Global Function score, an average of the 4 functional assessments, and a Happiness score are calculated. Normative scores are calculated so that higher scores indicate better functioning. All scores are referenced to the general, healthy population with a normative mean score of 50 and a standard deviation of 10. Population: one participant in the "Burosumab Q4W then Q2W" group did not have a Baseline assessment
  T-score
    Upper Extremity Scale: number analyzed (Participants) | 26 | 25 | 51
    Upper Extremity Scale | 52.1 (6.77) | 48.5 (13.04) | 50.3 (10.39)
    Transfer and Basic Mobility Scale: number analyzed (Participants) | 26 | 25 | 51
    Transfer and Basic Mobility Scale | 45.7 (10.88) | 46.0 (10.53) | 45.8 (10.61)
    Sports/Physical Functioning Scale: number analyzed (Participants) | 26 | 25 | 51
    Sports/Physical Functioning Scale | 34.6 (15.70) | 32.2 (19.29) | 33.4 (17.42)
    Pain/Comfort Scale: number analyzed (Participants) | 26 | 25 | 51
    Pain/Comfort Scale | 35.2 (15.26) | 34.8 (16.76) | 35.0 (15.85)
    Happiness Scale: number analyzed (Participants) | 26 | 25 | 51
    Happiness Scale | 43.6 (13.75) | 43.4 (13.69) | 43.5 (13.58)
    Global Functioning Scale: number analyzed (Participants) | 26 | 25 | 51
    Global Functioning Scale | 37.5 (13.96) | 35.6 (17.24) | 36.6 (15.52)
Fractional Excretion of Phosphorus (FEP) [Mean (Standard Deviation); unit: percentage of phosphorus excreted] — FEP is defined as 100% × (urine phosphorus × serum creatinine)/(urine creatinine × serum phosphorus), where the 2-hour urine sample was used for urine phosphorus and urine creatinine. Population: participants with a Baseline assessment
  percentage of phosphorus excreted
    number analyzed (Participants) | 25 | 26 | 51
    (all) | 13.91 (6.775) | 15.42 (7.373) | 14.68 (7.056)
Procollagen Type 1 N Propeptide (P1NP) [Mean (Standard Deviation); unit: ng/mL] — Population: participants with a Baseline assessment
  ng/mL
    number analyzed (Participants) | 24 | 26 | 50
    (all) | 843.11 (214.367) | 742.35 (209.727) | 790.72 (215.864)
Carboxy-Terminal Crosslinked Telopeptide of Type I Collagen (CTx) [Mean (Standard Deviation); unit: ng/mL] | 2.23 (0.642) | 2.10 (0.679) | 2.16 (0.658)
Alkaline Phosphatase (ALP) [Mean (Standard Deviation); unit: U/L] | 461.92 (110.209) | 456.08 (101.157) | 459.00 (104.779)
Bone Specific Alkaline Phosphatase (BALP) [Mean (Standard Deviation); unit: mcg/L] — Population: participants with a baseline assessment
  mcg/L
    number analyzed (Participants) | 20 | 20 | 40
    (all) | 163.54 (58.610) | 165.62 (45.534) | 164.58 (51.814)
Burosumab Concentration [Mean (Standard Deviation); unit: ng/mL] — For the lower limit of quantitation (< 50), the value 25 was used.
  ng/mL | 25.00 (0.000) | 25.00 (0.000) | 25.00 (0.000)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in RSS Total Score Over Time
Description: The RSS system is a 10-point radiographic scoring method that was developed to assess the severity of nutritional rickets in the wrists and knees based on the degree of metaphyseal fraying, cupping, and the proportion of the growth plate affected. Scores are assigned for the unilateral wrist and knee X-rays deemed by the rater to be the more severe of the bilateral images. The maximum total score on the RSS is 10 points and the minimum score is 0, with a total possible score of 4 points for the wrists and 6 points for the knees. Higher scores indicate greater rickets severity.
Time Frame: Baseline, Week 40, 64, 160
Population: Intent to Treat (ITT) Analysis Set: all participants who received at least 1 dose of study therapy and had at least 1 post-dose measurement at given time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Burosumab Q2W: Burosumab SC injections Q2W. Dose was determined by the participant's weight and prescribed dose by their study doctor.
- Burosumab Q4W Then Q2W: Burosumab SC injections Q4W. Dose was determined by the participant's weight and prescribed dose by their study doctor. Participants in Q4W were to switch to Q2W beginning with Week 64 dosing.
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 26
score on a scale
  Change to Week 40 | -1.06 (0.100) | -0.73 (0.100)
  Change to Week 64 | -1.00 (0.110) | -0.84 (0.098)
  Change to Week 160: number analyzed (Participants) | 19 | 22
  Change to Week 160 | -0.98 (0.129) | -0.83 (0.122)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 40; Test type: Superiority; p < 0.0001, GEE model — Per generalized estimating equations (GEE) model, which included visit, regimen, visit by regimen as factors, and RSS total score at baseline as a covariate, with exchangeable covariance structure
Statistical Analysis 2: Comparison: Burosumab Q4W Then Q2W; Week 40; Test type: Superiority; p < 0.0001, GEE model — Per GEE model, which included visit, regimen, visit by regimen as factors, and RSS total score at baseline as a covariate, with exchangeable covariance structure
Statistical Analysis 3: Comparison: Burosumab Q2W vs Burosumab Q4W Then Q2W; Difference in change to Week 40; Test type: Superiority; Difference in LS Means = -0.33, 95% CI 2-sided [-0.63 to -0.04]
Statistical Analysis 4: Comparison: Burosumab Q2W; Week 64; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Burosumab Q4W Then Q2W; Week 64; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Burosumab Q2W vs Burosumab Q4W Then Q2W; Difference in change to Week 64; Test type: Superiority; Difference in LS Means = -0.16, 95% CI 2-sided [-0.45 to 0.13]
Statistical Analysis 7: Comparison: Burosumab Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Burosumab Q4W Then Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 1, analysis 2]

2. Primary Outcome: Change From Baseline in Serum Phosphorus Over Time
Time Frame: Baseline, Week 40, 64, 160
Population: Pharmacokinetic/Pharamcodynamic (PK/PD) Analysis Set: all participants who received at least 1 dose of therapy and had evaluable serum data at given time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 26
mg/dL
  Change at Week 40 | 0.92 (0.480) | 0.57 (0.265)
  Change at Week 64: number analyzed (Participants) | 24 | 23
  Change at Week 64 | 0.99 (0.502) | 0.69 (0.370)
  Change at Week 160 | 0.97 (0.338) | 1.08 (0.377)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 40; Test type: Superiority; p < 0.0001, one sample t test
Statistical Analysis 2: Comparison: Burosumab Q4W Then Q2W; Week 40; Test type: Superiority; p < 0.0001, one sample t test
Statistical Analysis 3: Comparison: Burosumab Q2W; Week 64; Test type: Superiority; p < 0.0001, one sample t test
Statistical Analysis 4: Comparison: Burosumab Q4W Then Q2W; Week 64; Test type: Superiority; p < 0.0001, one sample t test
Statistical Analysis 5: Comparison: Burosumab Q2W; Week 160; Test type: Superiority; p < 0.0001, one sample t test
Statistical Analysis 6: Comparison: Burosumab Q4W Then Q2W; Week 160; Test type: Superiority; p < 0.0001, one sample t test

3. Primary Outcome: Change From Baseline in Serum 1,25(OH)2D Over Time
Time Frame: Baseline, Week 40, 64, 160
Population: PK/PD Analysis Set: all participants who received at least 1 dose of therapy and had evaluable serum data at given time point.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 26
pg/mL
  Change at Week 40 | 28.27 (29.312) | 17.62 (18.802)
  Change at Week 64: number analyzed (Participants) | 26 | 24
  Change at Week 64 | 23.58 (24.502) | 11.50 (16.522)
  Change at Week 160 | 17.03 (24.889) | 19.64 (22.857)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 40; Test type: Superiority; p < 0.0001, one sample t test
Statistical Analysis 2: Comparison: Burosumab Q4W Then Q2W; Week 40; Test type: Superiority; p < 0.0001, one sample t test
Statistical Analysis 3: Comparison: Burosumab Q2W; Week 64; Test type: Superiority; p < 0.0001, one sample t test
Statistical Analysis 4: Comparison: Burosumab Q4W Then Q2W; Week 64; Test type: Superiority; p = 0.0024, one sample t test
Statistical Analysis 5: Comparison: Burosumab Q2W; Week 160; Test type: Superiority; p = 0.0018, one sample t test
Statistical Analysis 6: Comparison: Burosumab Q4W Then Q2W; Week 160; Test type: Superiority; p = 0.0002, one sample t test

4. Primary Outcome: Change From Baseline in TmP/GFR Over Time
Description: Data for urinary phosphorus and TRP were used in calculation TmP/GFR.
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 26
mg/dL
  Change at Week 40: number analyzed (Participants) | 24 | 23
  Change at Week 40 | 1.14 (0.686) | 0.80 (0.506)
  Change at Week 64: number analyzed (Participants) | 20 | 19
  Change at Week 64 | 1.11 (0.626) | 0.90 (0.632)
  Change at Week 160: number analyzed (Participants) | 23 | 24
  Change at Week 160 | 1.24 (0.548) | 1.45 (0.653)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 40; Test type: Superiority; p < 0.0001, one sample t test
Statistical Analysis 2: Comparison: Burosumab Q4W Then Q2W; Week 40; Test type: Superiority; p < 0.0001, one sample t test
Statistical Analysis 3: Comparison: Burosumab Q2W; Week 64; Test type: Superiority; p < 0.0001, one sample t test
Statistical Analysis 4: Comparison: Burosumab Q4W Then Q2W; Week 64; Test type: Superiority; p < 0.0001, one sample t test
Statistical Analysis 5: Comparison: Burosumab Q2W; Week 160; Test type: Superiority; p < 0.0001, one sample t test
Statistical Analysis 6: Comparison: Burosumab Q4W Then Q2W; Week 160; Test type: Superiority; p < 0.0001, one sample t test

5. Secondary Outcome: Change From Baseline in RSS Knee Scores Over Time
Description: as for outcome 1
Time Frame: Baseline, Week 40, 64, 160
Population: ITT Analysis Set: all participants who received at least 1 dose of study therapy and had at least 1 post-dose measurement at given time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 26
score on a scale
  Change at Week 40 | -0.62 (0.08) | -0.55 (0.08)
  Change at Week 64 | -0.70 (0.087) | -0.61 (0.072)
  Change at Week 160: number analyzed (Participants) | 19 | 22
  Change at Week 160 | -0.70 (0.105) | -0.62 (0.093)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 40; Test type: Superiority; p < 0.0001, ANCOVA — ANCOVA model includes the change from baseline in RSS as the dependent variable, regimen group as factor, and RSS at baseline as covariate
Statistical Analysis 2: Comparison: Burosumab Q4W Then Q2W; Week 40; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Burosumab Q2W; Week 64; Test type: Superiority; p < 0.0001, GEE model — GEE model includes the change from baseline in RSS as the dependent variable, visit, regimen, visit by regimen as factors, and RSS at baseline as a covariate, with exchangeable covariance structure
Statistical Analysis 4: Comparison: Burosumab Q4W Then Q2W; Week 64; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 5, analysis 3]
Statistical Analysis 5: Comparison: Burosumab Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 5, analysis 3]
Statistical Analysis 6: Comparison: Burosumab Q4W Then Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 5, analysis 3]

6. Secondary Outcome: Change From Baseline in RSS Wrist Scores Over Time
Description: as for outcome 1
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 26
score on a scale
  Change at Week 40 | -0.44 (0.05) | -0.18 (0.05)
  Change at Week 64 | -0.30 (0.057) | -0.24 (0.051)
  Change at Week 160: number analyzed (Participants) | 19 | 21
  Change at Week 160 | -0.27 (0.065) | -0.20 (0.047)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 40; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Burosumab Q4W Then Q2W; Week 40; Test type: Superiority; p = 0.0015, ANCOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Burosumab Q2W; Week 64; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 5, analysis 3]
Statistical Analysis 4: Comparison: Burosumab Q4W Then Q2W; Week 64; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 5, analysis 3]
Statistical Analysis 5: Comparison: Burosumab Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 5, analysis 3]
Statistical Analysis 6: Comparison: Burosumab Q4W Then Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 5, analysis 3]

7. Secondary Outcome: Radiographic Global Impression of Change (RGI-C) Global Scores Over Time
Description: Changes in the severity of rickets and bowing were assessed centrally by three independent pediatric radiologists contracted by a central imaging facility using a disease specific qualitative RGI-C scoring system. The RGI-C is a seven point ordinal scale with possible values: +3 = very much better (complete or near complete healing of rickets), +2 = much better (substantial healing of rickets), +1 = minimally better (i.e., minimal healing of rickets), 0 = unchanged, -1 = minimally worse (minimal worsening of rickets), -2 = much worse (moderate worsening of rickets), -3 = very much worse (severe worsening of rickets).
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 26
score on a scale
  Change at Week 40 | 1.67 (0.12) | 1.46 (0.12)
  Change at Week 64 | 1.56 (0.112) | 1.58 (0.112)
  Change at Week 160 | 1.92 (0.111) | 1.86 (0.119)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 40; Test type: Superiority; p < 0.0001, ANCOVA — ANCOVA model includes RGI-C as the dependent variable, regimen group as factor, and RSS at baseline as covariate
Statistical Analysis 2: Comparison: Burosumab Q4W Then Q2W; Week 40; Test type: Superiority; p < 0.0001, ANCOVA — ANCOVA model includes RGI-C as the dependent variable, regimen group as factor, and RSS at baseline as covariate
Statistical Analysis 3: Comparison: Burosumab Q2W vs Burosumab Q4W Then Q2W; Difference in change to Week 40; Test type: Superiority; Difference in LS Means = 0.21, 95% CI 2-sided [-0.12 to 0.54]
Statistical Analysis 4: Comparison: Burosumab Q2W; Week 64; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Burosumab Q4W Then Q2W; Week 64; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Burosumab Q2W vs Burosumab Q4W Then Q2W; Difference in change to Week 64; Test type: Superiority; Difference in LS Means = -0.02, 95% CI 2-sided [-0.34 to 0.29]
Statistical Analysis 7: Comparison: Burosumab Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Burosumab Q4W Then Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 1, analysis 2]

8. Secondary Outcome: RGI-C Knee Scores Over Time
Description: as for outcome 7
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 26
score on a scale
  Change at Week 40 | 1.60 (0.13) | 1.34 (0.13)
  Change at Week 64 | 1.57 (0.104) | 1.53 (0.099)
  Change at Week 160 | 2.01 (0.106) | 1.85 (0.118)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 40; Test type: Superiority; p < 0.0001, ANCOVA — ANCOVA model includes RGI-C as the dependent variable, regimen group as factor, and RSS at baseline as covariate
Statistical Analysis 2: Comparison: Burosumab Q4W Then Q2W; Week 40; Test type: Superiority; p < 0.0001, ANCOVA — ANCOVA model includes RGI-C as the dependent variable, regimen group as factor, and RSS at baseline as covariate
Statistical Analysis 3: Comparison: Burosumab Q2W; Week 64; Test type: Superiority; p < 0.0001, GEE model — GEE model includes RGI-C as the dependent variable, visit, regimen, visit by regimen as factors, and RSS total score at baseline as a covariate, with exchangeable covariance structure
Statistical Analysis 4: Comparison: Burosumab Q4W Then Q2W; Week 64; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 8, analysis 3]
Statistical Analysis 5: Comparison: Burosumab Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 8, analysis 3]
Statistical Analysis 6: Comparison: Burosumab Q4W Then Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 8, analysis 3]

9. Secondary Outcome: RGI-C Wrist Scores Over Time
Description: as for outcome 7
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 26
score on a scale
  Change at Week 40 | 1.64 (0.14) | 1.45 (0.14)
  Change at Week 64 | 1.65 (0.153) | 1.55 (0.124)
  Change at Week 160: number analyzed (Participants) | 26 | 25
  Change at Week 160 | 1.78 (0.133) | 1.83 (0.132)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 40; Test type: Superiority; p < 0.0001, ANCOVA — ANCOVA model includes RGI-C as the dependent variable, regimen group as factor, and RSS at baseline as covariate
Statistical Analysis 2: Comparison: Burosumab Q4W Then Q2W; Week 40; Test type: Superiority; p < 0.0001, ANCOVA — ANCOVA model includes RGI-C as the dependent variable, regimen group as factor, and RSS at baseline as covariate
Statistical Analysis 3: Comparison: Burosumab Q2W; Week 64; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 8, analysis 3]
Statistical Analysis 4: Comparison: Burosumab Q4W Then Q2W; Week 64; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 8, analysis 3]
Statistical Analysis 5: Comparison: Burosumab Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 8, analysis 3]
Statistical Analysis 6: Comparison: Burosumab Q4W Then Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 8, analysis 3]

10. Secondary Outcome: Change From Baseline in Growth Velocity Over Time
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 25 | 24
cm/year
  Week 0 to Week 40: Change from Baseline | 0.96 (1.677) | 0.39 (2.559)
  Week 0 to Week 64: Change from Baseline | 0.73 (1.399) | 0.37 (2.164)
  Week 64 to Week 112: Change from Baseline | 0.29 (2.284) | 0.09 (2.523)
  Week 112 to Week 160: Change from Baseline | 0.67 (2.318) | 0.54 (3.158)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 0 to Week 40; Test type: Superiority; p = 0.0088, one sample t-test
Statistical Analysis 2: Comparison: Burosumab Q4W Then Q2W; Week 0 to Week 40; Test type: Superiority; p = 0.4650, one sample t-test
Statistical Analysis 3: Comparison: Burosumab Q2W; Week 0 to Week 64; Test type: Superiority; p = 0.0160, one sample t test
Statistical Analysis 4: Comparison: Burosumab Q4W Then Q2W; Week 0 to Week 64; Test type: Superiority; p = 0.4114, one sample t test
Statistical Analysis 5: Comparison: Burosumab Q2W; Week 64 to Week 112; Test type: Superiority; p = 0.5335, one sample t test
Statistical Analysis 6: Comparison: Burosumab Q4W Then Q2W; Week 64 to Week 112; Test type: Superiority; p = 0.8606, one sample t test
Statistical Analysis 7: Comparison: Burosumab Q2W; Week 112 to Week 160; Test type: Superiority; p = 0.1627, one sample t test
Statistical Analysis 8: Comparison: Burosumab Q4W Then Q2W; Week 112 to Week 160; Test type: Superiority; p = 0.4096, one sample t test

11. Secondary Outcome: Change From Baseline in Standing Height Z Score Over Time
Description: Standing height Z scores are measures of height adjusted for a child's age and sex. The Z score indicates the number of standard deviations away from a reference population (from the CDC growth charts) in the same age range and with the same sex. A Z score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z scores indicate a better outcome.
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Z score
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 26
Z score
  Change to Week 40: number analyzed (Participants) | 24 | 23
  Change to Week 40 | 0.17 (0.042) | 0.10 (0.051)
  Change to Week 64 | 0.19 (0.051) | 0.12 (0.061)
  Change to Week 160 | 0.35 (0.084) | 0.19 (0.089)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 40; Test type: Superiority; p < 0.0001, GEE model — GEE model included change from baseline for standing height Z score as dependent variable; visit, regimen, visit by regimen, and gender as factors; and age and standing height Z score at baseline as covariates, with exchangeable covariance structure
Statistical Analysis 2: Comparison: Burosumab Q4W Then Q2W; Week 40; Test type: Superiority; p = 0.0569, GEE model — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Burosumab Q2W; Week 64; Test type: Superiority; p = 0.0002, GEE model — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 4: Comparison: Burosumab Q4W Then Q2W; Week 64; Test type: Superiority; p = 0.0456, GEE model — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 5: Comparison: Burosumab Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 11, analysis 1]
Statistical Analysis 6: Comparison: Burosumab Q4W Then Q2W; Week 160; Test type: Superiority; p = 0.0343, GEE model — [p-value comment as in outcome 11, analysis 1]

12. Secondary Outcome: Change From Baseline in Growth (Standing Height) Over Time
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 26
cm
  Change at Week 40: number analyzed (Participants) | 24 | 23
  Change at Week 40 | 5.03 (1.232) | 4.49 (1.455)
  Change at Week 64 | 7.48 (1.934) | 6.98 (1.594)
  Change at Week 160 | 18.38 (2.958) | 17.22 (2.653)

13. Secondary Outcome: Change From Baseline in Growth (Sitting Height) Over Time
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 26
cm
  Change at Week 40: number analyzed (Participants) | 23 | 23
  Change at Week 40 | 2.66 (5.496) | 2.39 (1.486)
  Change at Week 64 | 3.08 (2.405) | 3.45 (1.390)
  Change at Week 160 | 8.29 (2.928) | 8.62 (2.163)

14. Secondary Outcome: Change From Baseline in Growth (Arm Length) Over Time
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 26
cm
  Change at Week 40: number analyzed (Participants) | 24 | 23
  Change at Week 40 | 2.36 (1.058) | 2.08 (0.905)
  Change at Week 64 | 3.99 (1.556) | 4.77 (7.382)
  Change at Week 160 | 8.50 (1.537) | 8.32 (1.798)

15. Secondary Outcome: Change From Baseline in Growth (Leg Length) Over Time
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 26
cm
  Change to Week 40: number analyzed (Participants) | 24 | 23
  Change to Week 40 | 2.90 (1.365) | 2.82 (1.270)
  Change at Week 64 | 5.03 (1.879) | 5.16 (1.283)
  Change at Week 160 | 11.78 (3.040) | 11.67 (2.338)

16. Secondary Outcome: 6MWT Distance (Predicted Percent of Normal) Change From Baseline Over Time
Description: The total distance walked (meters) in a 6-minute period was measured. The percent of predicted values were calculated using published normative data based on age, gender, and height (Geiger et al. 2007).
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percentage of predicted distance
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 26
percentage of predicted distance
  Change to Week 40 | 3.25 (1.841) | 0.24 (2.153)
  Change to Week 64 | 5.29 (1.568) | 3.70 (1.731)
  Change to Week 160 | 1.96 (1.483) | 2.15 (1.932)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 40; Test type: Superiority; p = 0.0771, GEE model — GEE model included change in 6MWT score as the dependent variable; visit, regimen, visit by regimen as factors; and 6MWT at baseline as a covariate, with exchangeable covariance structure
Statistical Analysis 2: Comparison: Burosumab Q4W Then Q2W; Week 40; Test type: Superiority; p = 0.9098, GEE model — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 3: Comparison: Burosumab Q2W; Week 64; Test type: Superiority; p = 0.0007, GEE model — GEE model included change in percent of predicted 6MWT score as the dependent variable; visit, regimen, visit by regimen as factors; and 6MWT at baseline as a covariate, with exchangeable covariance structure
Statistical Analysis 4: Comparison: Burosumab Q4W Then Q2W; Week 64; Test type: Superiority; p = 0.0327, GEE model — [p-value comment as in outcome 16, analysis 3]
Statistical Analysis 5: Comparison: Burosumab Q2W; Week 160; Test type: Superiority; p = 0.1865, GEE model — [p-value comment as in outcome 16, analysis 3]
Statistical Analysis 6: Comparison: Burosumab Q4W Then Q2W; Week 160; Test type: Superiority; p = 0.2654, GEE model — [p-value comment as in outcome 16, analysis 3]

17. Secondary Outcome: Change From Baseline in POSNA-PODCI (Normative Score) Upper Extremity Scale Scores Over Time
Description: The POSNA-PODCI yields 4 functional assessment scores: Upper Extremity Function,Transfers and Basic Mobility, Sports and Physical Function, and Comfort/Pain. In addition, a Global Function score, which is an average of the 4 functional assessments, and a Happiness score are calculated. Raw, mean, standardized, and normative scores are calculated for each scale. Normative scores are calculated so that higher scores indicate better functioning. All scores are referenced to the general, healthy population with a normative mean score of 50 and a standard deviation of 10.
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 25
T-score
  Change at Week 40: number analyzed (Participants) | 25 | 24
  Change at Week 40 | 2.97 (0.710) | 2.97 (1.212)
  Change at Week 64 | 1.89 (0.914) | 3.20 (0.911)
  Change at Week 160 | -0.02 (0.740) | 1.82 (1.449)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 40; Test type: Superiority; p < 0.0001, GEE model — GEE model includes change in POSNA-PODCI score as the dependent variable, visit, regimen, visit by regimen as factors, and POSNA-PODCI at baseline as a covariate, with exchangeable covariance structure
Statistical Analysis 2: Comparison: Burosumab Q4W Then Q2W; Week 40; Test type: Superiority; p = 0.0144, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 3: Comparison: Burosumab Q2W; Week 64; Test type: Superiority; p = 0.0384, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 4: Comparison: Burosumab Q4W Then Q2W; Week 64; Test type: Superiority; p = 0.0004, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 5: Comparison: Burosumab Q2W; Week 160; Test type: Superiority; p = 0.9795, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 6: Comparison: Burosumab Q4W Then Q2W; Week 160; Test type: Superiority; p = 0.2082, GEE model — [p-value comment as in outcome 17, analysis 1]

18. Secondary Outcome: Change From Baseline in POSNA-PODCI (Normative Score) Transfer and Basic Mobility Scale Scores Over Time
Description: as for outcome 17
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 25
T-score
  Change at Week 40: number analyzed (Participants) | 25 | 24
  Change at Week 40 | 4.04 (0.827) | 3.69 (1.648)
  Change at Week 64 | -0.34 (3.123) | 4.32 (1.364)
  Change at Week 160 | 1.88 (3.285) | 5.44 (1.113)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 40; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 2: Comparison: Burosumab Q4W Then Q2W; Week 40; Test type: Superiority; p = 0.0251, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 3: Comparison: Burosumab Q2W; Week 64; Test type: Superiority; p = 0.9124, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 4: Comparison: Burosumab Q4W Then Q2W; Week 64; Test type: Superiority; p = 0.0016, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 5: Comparison: Burosumab Q2W; Week 160; Test type: Superiority; p = 0.5677, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 6: Comparison: Burosumab Q4W Then Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 17, analysis 1]

19. Secondary Outcome: Change From Baseline in POSNA-PODCI (Normative Score) Sports/Physical Functioning Scale Scores Over Time
Description: as for outcome 17
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 25
T-score
  Change at Week 40: number analyzed (Participants) | 25 | 24
  Change at Week 40 | 9.78 (1.679) | 9.15 (2.249)
  Change at Week 64 | 7.74 (2.636) | 9.84 (2.534)
  Change at Week 160: number analyzed (Participants) | 25 | 25
  Change at Week 160 | 12.04 (2.102) | 14.33 (1.834)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 40; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 2: Comparison: Burosumab Q4W Then Q2W; Week 40; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 3: Comparison: Burosumab Q2W; Week 64; Test type: Superiority; p = 0.0033, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 4: Comparison: Burosumab Q4W Then Q2W; Week 64; Test type: Superiority; p = 0.0001, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 5: Comparison: Burosumab Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 6: Comparison: Burosumab Q4W Then Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 17, analysis 1]

20. Secondary Outcome: Change From Baseline in POSNA-PODCI (Normative Score) Pain/Comfort Scale Scores Over Time
Description: as for outcome 17
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 25
T-score
  Change at Week 40: number analyzed (Participants) | 25 | 24
  Change at Week 40 | 7.67 (2.399) | 7.39 (2.477)
  Change at Week 64 | 5.60 (2.904) | 7.74 (2.077)
  Change at Week 160 | 13.06 (2.187) | 12.38 (2.265)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 40; Test type: Superiority; p = 0.0014, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 2: Comparison: Burosumab Q4W Then Q2W; Week 40; Test type: Superiority; p = 0.0028, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 3: Comparison: Burosumab Q2W; Week 64; Test type: Superiority; p = 0.0536, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 4: Comparison: Burosumab Q4W Then Q2W; Week 64; Test type: Superiority; p = 0.0002, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 5: Comparison: Burosumab Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 6: Comparison: Burosumab Q4W Then Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 17, analysis 1]

21. Secondary Outcome: Change From Baseline in POSNA-PODCI (Normative Score) Happiness Scale Scores Over Time
Description: as for outcome 17
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 25
T-score
  Change at Week 40: number analyzed (Participants) | 25 | 24
  Change at Week 40 | 2.84 (2.328) | 3.01 (1.902)
  Change at Week 64 | 2.18 (1.914) | 3.34 (1.914)
  Change at Week 160 | 6.46 (2.486) | 9.19 (1.075)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 40; Test type: Superiority; p = 0.2230, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 2: Comparison: Burosumab Q4W Then Q2W; Week 40; Test type: Superiority; p = 0.1132, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 3: Comparison: Burosumab Q2W; Week 64; Test type: Superiority; p = 0.2558, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 4: Comparison: Burosumab Q4W Then Q2W; Week 64; Test type: Superiority; p = 0.0814, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 5: Comparison: Burosumab Q2W; Week 160; Test type: Superiority; p = 0.0093, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 6: Comparison: Burosumab Q4W Then Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 17, analysis 1]

22. Secondary Outcome: Change From Baseline in POSNA-PODCI (Normative Score) Global Functioning Scale Scores Over Time
Description: as for outcome 17
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 25
T-score
  Change at Week 40: number analyzed (Participants) | 25 | 24
  Change at Week 40 | 9.06 (1.560) | 8.12 (2.351)
  Change at Week 64 | 6.02 (2.706) | 8.72 (2.019)
  Change at Week 160: number analyzed (Participants) | 25 | 25
  Change at Week 160 | 11.37 (1.804) | 11.94 (2.024)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 40; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 2: Comparison: Burosumab Q4W Then Q2W; Week 40; Test type: Superiority; p = 0.0006, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 3: Comparison: Burosumab Q2W; Week 64; Test type: Superiority; p = 0.0260, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 4: Comparison: Burosumab Q4W Then Q2W; Week 64; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 5: Comparison: Burosumab Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 17, analysis 1]
Statistical Analysis 6: Comparison: Burosumab Q4W Then Q2W; Week 160; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 17, analysis 1]

23. Secondary Outcome: Change From Baseline in FEP Over Time
Description: FEP is defined as 100% × (urine phosphorus × serum creatinine)/(urine creatinine × serum phosphorus), where the 2-hour urine sample was used for urine phosphorus and urine creatinine.
Time Frame: Baseline, Week 40, 64, 160
Population: Safety Analysis Set: All participants who received at least 1 dose of study therapy and had an assessment at given time point.
Measure: Mean (Standard Deviation); unit: percentage of phosphorus excreted
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 25 | 26
percentage of phosphorus excreted
  Change at Week 40 | -3.97 (7.161) | -4.85 (7.170)
  Change at Week 64: number analyzed (Participants) | 20 | 22
  Change at Week 64 | -2.63 (4.446) | -3.96 (7.522)
  Change at Week 160: number analyzed (Participants) | 23 | 26
  Change at Week 160 | -5.43 (6.985) | -6.47 (8.072)

24. Secondary Outcome: Change From Baseline in P1NP Over Time
Time Frame: Baseline, Week 40, 64
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 24 | 26
ng/mL
  Change at Week 40 | 275.98 (329.587) | 224.91 (161.053)
  Change at Week 64: number analyzed (Participants) | 22 | 23
  Change at Week 64 | 137.35 (354.315) | 133.56 (192.306)

25. Secondary Outcome: Change From Baseline in CTx Over Time
Time Frame: Baseline, Week 40, 64
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 26
ng/mL
  Change at Week 40 | 1.01 (0.802) | 0.64 (0.578)
  Change at Week 64: number analyzed (Participants) | 25 | 25
  Change at Week 64 | 1.08 (0.870) | 0.81 (0.706)

26. Secondary Outcome: Change From Baseline in ALP Over Time
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 26
U/L
  Change at Week 40 | -79.4 (97.40) | -47.8 (70.86)
  Change at Week 64: number analyzed (Participants) | 24 | 23
  Change at Week 64 | -113.9 (81.28) | -80.9 (67.11)
  Change at Week 160 | -153.1 (132.45) | -140.0 (115.82)
Statistical Analysis 1: Comparison: Burosumab Q2W; Week 40; Test type: Superiority; p = 0.0003, one sample t test
Statistical Analysis 2: Comparison: Burosumab Q4W Then Q2W; Week 40; Test type: Superiority; p = 0.0021, one sample t test
Statistical Analysis 3: Comparison: Burosumab Q2W; Week 64; Test type: Superiority; p < 0.0001, one sample t test
Statistical Analysis 4: Comparison: Burosumab Q4W Then Q2W; Week 64; Test type: Superiority; p < 0.0001, one sample t test
Statistical Analysis 5: Comparison: Burosumab Q2W; Week 160; Test type: Superiority; p < 0.0001, one sample t test
Statistical Analysis 6: Comparison: Burosumab Q4W Then Q2W; Week 160; Test type: Superiority; p < 0.0001, one sample t test

27. Secondary Outcome: Change From Baseline in BALP Over Time
Time Frame: Baseline, Week 40, 64, 160
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 20 | 20
mcg/L
  Change at Week 40 | -35.55 (46.738) | -27.80 (31.409)
  Change at Week 64: number analyzed (Participants) | 19 | 20
  Change at Week 64 | -50.40 (36.478) | -47.13 (28.822)
  Change at Week 160 | -67.25 (59.309) | -56.73 (52.284)

28. Secondary Outcome: Serum Pre-Dose Concentrations of Burosumab
Time Frame: Week 40, 64, 160
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 26
ng/mL
  Week 40 | 13188.81 (7188.588) | 6443.08 (3266.215)
  Week 64: number analyzed (Participants) | 26 | 24
  Week 64 | 15846.65 (9385.393) | 8525.63 (3968.821)
  Week 160 | 13975.27 (8168.877) | 13163.96 (6593.120)

29. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Discontinuations Due to Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An SAE is defined as an AE or suspected adverse reaction that at any dose results in any of the following outcomes: death; life-threatening AE; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; a congenital anomaly/birth defect. Severity was graded as 1 (mild), 2 (moderate), 3 (severe), 4 (life-threatening), 5 (death). TEAEs are defined as AEs with onset on or after the time of initiation of study drug administration.
Time Frame: Up to 216 weeks
Population: Safety Analysis Set: All participants who received at least 1 dose of study therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
Number analyzed (Participants) | 26 | 26
Participants
  All TEAEs | 26 | 26
  Serious TEAE | 0 | 1
  Related TEAE | 17 | 21
  Serious Related TEAE | 0 | 1
  Grade 3 or 4 TEAE | 1 | 1
  TEAE Leading to Study Discontinuation | 0 | 0
  TEAE Leading to Treatment Discontinuation | 0 | 0
  TEAE Leading to Death | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 216 weeks
Description: TEAEs, defined as AEs with onset on or after the time of initiation of study drug administration, are presented.
Arm/Group | Burosumab Q2W | Burosumab Q4W Then Q2W
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 1/26
Other Adverse Events (participants affected / at risk) | 26/26 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Burosumab Q2W (N=26) | Burosumab Q4W Then Q2W (N=26)
Pyrexia (General disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Burosumab Q2W (N=26) | Burosumab Q4W Then Q2W (N=26)
Ear Pain (Ear and labyrinth disorders) | 10 | 8
Dry Eye (Eye disorders) | 0 | 3
Eye Pain (Eye disorders) | 2 | 2
Eye Pruritus (Eye disorders) | 3 | 2
Lacrimation Increased (Eye disorders) | 1 | 3
Abdominal Discomfort (Gastrointestinal disorders) | 4 | 2
Abdominal Pain (Gastrointestinal disorders) | 2 | 7
Abdominal Pain Upper (Gastrointestinal disorders) | 10 | 8
Constipation (Gastrointestinal disorders) | 2 | 4
Dental Caries (Gastrointestinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 7 | 11
Gingival Pain (Gastrointestinal disorders) | 0 | 2
Lip Swelling (Gastrointestinal disorders) | 0 | 2
Mouth Ulceration (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 9 | 8
Oral Pain (Gastrointestinal disorders) | 2 | 3
Toothache (Gastrointestinal disorders) | 6 | 11
Vomiting (Gastrointestinal disorders) | 13 | 16
Fatigue (General disorders) | 5 | 3
Influenza Like Illness (General disorders) | 2 | 1
Injection Site Bruising (General disorders) | 5 | 4
Injection Site Erythema (General disorders) | 14 | 9
Injection Site Pain (General disorders) | 3 | 3
Injection Site Pruritus (General disorders) | 2 | 4
Injection Site Rash (General disorders) | 2 | 2
Injection Site Reaction (General disorders) | 13 | 13
Injection Site Swelling (General disorders) | 5 | 1
Malaise (General disorders) | 3 | 3
Medical Device Pain (General disorders) | 3 | 2
Non-Cardiac Chest Pain (General disorders) | 0 | 2
Pain (General disorders) | 6 | 4
Peripheral Swelling (General disorders) | 1 | 2
Pyrexia (General disorders) | 12 | 13
Seasonal Allergy (Immune system disorders) | 6 | 11
Conjunctivitis (Infections and infestations) | 3 | 0
Ear Infection (Infections and infestations) | 4 | 3
Enterobiasis (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 2 | 0
Gastroenteritis Viral (Infections and infestations) | 2 | 4
Gingival Abscess (Infections and infestations) | 1 | 2
Infectious Mononucleosis (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 6 | 4
Lice Infestation (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 13 | 15
Pharyngitis Streptococcal (Infections and infestations) | 4 | 6
Rhinitis (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 3 | 3
Tooth Abscess (Infections and infestations) | 3 | 6
Upper Respiratory Tract Infection (Infections and infestations) | 12 | 13
Viral Infection (Infections and infestations) | 3 | 2
Viral Upper Respiratory Tract Infection (Infections and infestations) | 5 | 3
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 6 | 5
Fall (Injury, poisoning and procedural complications) | 3 | 3
Joint Injury (Injury, poisoning and procedural complications) | 2 | 2
Laceration (Injury, poisoning and procedural complications) | 2 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 3 | 2
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 6
Skin Abrasion (Injury, poisoning and procedural complications) | 3 | 4
Thermal Burn (Injury, poisoning and procedural complications) | 3 | 0
Blood 1,25-Dihydroxycholecalciferol Increased (Investigations) | 0 | 2
Blood 25-Hydroxycholecalciferol Decreased (Investigations) | 2 | 1
Blood Parathyroid Hormone Increased (Investigations) | 1 | 2
Vitamin D Decreased (Investigations) | 6 | 5
Vitamin D Deficiency (Metabolism and nutrition disorders) | 4 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 17
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 7
Neck Pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 10 | 17
Scoliosis (Musculoskeletal and connective tissue disorders) | 3 | 1
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Dizziness (Nervous system disorders) | 2 | 7
Headache (Nervous system disorders) | 20 | 19
Lethargy (Nervous system disorders) | 1 | 2
Migraine (Nervous system disorders) | 5 | 1
Post-Traumatic Headache (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 3 | 0
Initial Insomnia (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 4 | 1
Glycosuria (Renal and urinary disorders) | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 1
Menorrhagia (Reproductive system and breast disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 14 | 12
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 12 | 10
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 4
Eczema (Skin and subcutaneous tissue disorders) | 1 | 3
Erythema (Skin and subcutaneous tissue disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 5
Rash (Skin and subcutaneous tissue disorders) | 7 | 8
Swelling Face (Skin and subcutaneous tissue disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT02163577/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT02163577/SAP_001.pdf